CLINICAL TRIAL: NCT06997900
Title: Menopur And Rekovelle Combination Study Version 2.0
Acronym: MARCS 2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-1056
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: IVF; Controlled Ovarian Simulation; Fertility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follitropin delta and HP-hMG (Experimental)
  Interventions: Drug: Combination therapy : Follitropin delta and HP-hMG

INTERVENTIONS:
Drug: Combination therapy : Follitropin delta and HP-hMG — Follitropin delta dose will be determined by age. Highly purified human menopausal gonadotrophin will be determined by follitropin delta dose and body weight.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of a personalized ovarian stimulation regimen in women aged 18 to 40 undergoing in vitro fertilization (IVF). The main question it aims to answer is:

- Does personalizing the starting doses of follitropin delta (REKOVELLE) and HP-hMG (MENOPUR) based on both age and body lead to similar results as anti-Müllerian hormone (AMH) and weight based dosing ?

Researchers will compare the new dosing regimen to the MARCS study results to see if this new approach leads to similar outcomes

Participants will:

* Receive ovarian stimulation using a personalized dose of REKOVELLE aND MENOPUR based on age and weight
* Be monitored through ultrasound imaging and blood tests to measure estradiol (E2) levels
* Undergo standard IVF procedures including egg retrieval and embryo assessment

DETAILED DESCRIPTION:
In vitro fertilization (IVF) is a multi-step process that includes controlled ovarian stimulation, oocyte retrieval, fertilization, and embryo transfer. Success in IVF largely depends on how the ovaries respond to stimulation using exogenous gonadotropins. Luteinizing hormone (LH) and follicle-stimulating hormone (FSH) are key to folliculogenesis and oocyte maturation, and are central to ovarian stimulation protocols. Physicians typically determine the appropriate stimulation regimen by considering clinical factors such as age, body weight, and ovarian reserve, and choosing the type and dose of gonadotropins accordingly. The combined use of FSH and LH, such as in protocols incorporating both recombinant FSH and human menopausal gonadotropin (hMG), has shown improvements in ART outcomes.

Among gonadotropins, follitropin delta (REKOVELLE) is a recombinant FSH with allowing for individualized dosing based on anti-Müllerian hormone (AMH) levels and body weight. The ESTHER-1 trial demonstrated its safety and efficacy when personalized using this algorithm. Furthermore, the MARCS study showed that combining REKOVELLE with highly purified hMG (MENOPUR) led to higher number of retrieved oocytes and improved blastulation rate compared to REKOVELLE alone.

However, in some regions, AMH is not routinely used to personalize FSH dosing. Other trials, such as RITA-1 and RITA-2, demonstrated the potential of adjusting REKOVELLE doses based solely on age and body weight. Inspired by these findings, this study seeks to evaluate dosing based on age and weight for combination therapy with REKOVELLE and MENOPUR.

This is a prospective, interventional, phase II clinical trial enrolling 200 participants across two fertility centers in Canada. The objective is to determine whether individualizing the starting doses of REKOVELLE and MENOPUR based on age and body weight results in similar clinical outcomes to those achieved when dosing is based on AMH and weight, as per the standard REKOVELLE dosing algorithm.

Unlike the original MARCS protocol, which used a fixed dose of REKOVELLE and variable MENOPUR, this study will apply an adjustable REKOVELLE dose and a fixed MENOPUR dose. The study aims to assess ovarian response, blastulation, embryo quality, pregnancy rates, and safety outcomes, particularly the risk of ovarian hyperstimulation syndrome (OHSS).

This research will contribute valuable data on the feasibility and effectiveness of an age- and weight-based dosing regimen for REKOVELLE and MENOPUR mixed protocol ovarian stimulation, especially in clinical environments where AMH measurement is less accessible.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 40 years inclusively at the time of consent form signature
* Diagnosis of unexplained infertility, tubal infertility, endometriosis stage I/II or male factor infertility
* Regular menstrual cycles of 24-35 days
* Presence of both ovaries
* Early follicular phase FSH serum concentration <10 IU/L measured between Day 2 and Day 5 of menstrual cycle within the previous 24 months
* First IVF/ICSI cycle
* IVF antagonist protocol prescribed
* Partner or donor ejaculated sperm (fresh or frozen) used for fertilization

Exclusion Criteria:

* Women undergoing oocyte donation
* Endometriosis stage III/IV
* High risk of OHSS (AMH ≥ 35 pmol/L)
* Body Mass Index (BMI) > 40 kg/m2 Protocol number: IIS-1056 MARCS 2.0 Study Version: 1.1 - Date : 14 APR 2025 Page 12 of 28
* Gynaecological haemorrhages of unknown aetiology
* History of recurrent miscarriages defined as ≥ 3 consecutive losses
* Renal or hepatic impairment
* Hypersensitivity to any active ingredient or excipients in follitropin delta and/or HP-hMG
* Tumours of hypothalamus or pituitary gland
* Ovarian enlargement or ovarian cyst not due to polycystic ovarian syndrome
* Current or history of ovarian, uterine or mammary carcinoma
* History of thrombophilia
* Use of hormonal preparations (except for 17β-estradiol, testosterone gel, DHEA and thyroid medication) during the last menstrual cycle
* Women participating in any other interventional research project

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
number of good quality (>3BB) or utilizable blastocysts per treatment cycle at day 5 or 6 of embryo culture | 5 to 6 days after egg retrieval (up to 1 to 2 months after enrollment)

SECONDARY OUTCOMES:
Safety profile of follitropin delta + HP-hMG mixed protocol | up to 15 days after egg retrieval
  Patient rate that will develop ovarian hyperstimulation syndrome (OHSS)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Ottawa fertility centre, Ottawa, Ontario
  - Clinique ovo, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bissonnette F, Minano Masip J, Kadoch IJ, Librach C, Sampalis J, Yuzpe A. Individualized ovarian stimulation for in vitro fertilization: a multicenter, open label, exploratory study with a mixed protocol of follitropin delta and highly purified human menopausal gonadotropin. Fertil Steril. 2021 Apr;115(4):991-1000. doi: 10.1016/j.fertnstert.2020.09.158. Epub 2020 Nov 30. PMID 33267959